CLINICAL TRIAL: NCT03465761
Title: A Clinical Trial to Evaluate the Safety and Efficacy of Staged Bilateral Exablate Treatment of Medication Refractory Essential Tremor
Brief Title: Staged Bilateral Exablate Treatment of Medication Refractory Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET003
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Essential Tremor
Keywords: MRgFUS; ExAblate; Bilateral Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExAblate 4000 System (Experimental): ExAblate treatment of Bilateral Essential Tremor
  Interventions: Device: ExAblate

INTERVENTIONS:
Device: ExAblate — Bilateral side treatment of Essential Tremor

SUMMARY:
The objective of this prospective, multi-site, single-arm, open-label study is to capture the safety and efficacy (outcome) of bilateral staged Exablate treatment in subjects with bilateral medication-refractory essential tremor (ET). The staged second procedure will be performed at least 9 months after the first side. The benefit of real-time feedback will allow the physician to maximize benefit without jeopardizing safety.

This study is designed as a prospective, open-label, single arm, multi-site study design.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who:

   1. previously underwent Exablate thalamotomy for their essential tremor in a clinical study or in a commercial procedure at least 9 months prior to enrolling in this study for contralateral Exablate thalamotomy
   2. Subjects who would benefit from a bilateral treatment for their essential tremor and would want to undergo a staged bilateral thalamotomy
2. All subjects must have a complete baseline CRST prior from first Exablate thalamotomy
3. Men and women age 22 years to 75 years of age.
4. Minimum score of 24 on MoCA or 20 on MMSE
5. Subjects who are able and willing to give consent and able to attend all study visits
6. Postural or intention tremor severity score of greater than or equal to 2 in the both upper extremities as measured by the CRST rating scale while on stable medication
7. Thalamus can be targeted by the Exablate device. The region must be apparent on MRI such that targeting can be performed.
8. Able to communicate sensations during the Exablate Thalamotomy treatment
9. Original (before first Exablate procedure) CRST score of 2 or above in any one of the items 16-23 from the Disability subsection of the CRST: speaking, feeding other than liquids, bringing liquids to mouth, hygiene, dressing, writing, working, and social activities.
10. Subjects on antidepressant medications must be stable for at least 3 months prior to procedure(i.e., no change in medication drug or dosage for 3 months based on historical medical records).
11. Remains eligible for Exablate treatment with no changes to medical history that would affect Exablate treatment criteria, (e.g., bleeding/coagulation requirements, or new pathology such as infarct, tumor, etc).

Exclusion Criteria:

1. Subjects with unstable cardiac status
2. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within a 12 month period:
3. Subjects with uncontrollable blood pressure (hypertensive with diastolic BP > 100 on medication)
4. History of abnormal bleeding and/or coagulopathy, i.e. subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard
5. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
6. Active or suspected acute or chronic uncontrolled infection
7. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
8. Subjects with life-threatening systemic disease that include but not limited to the following will be excluded from the study participation: HIV, Liver Failure, blood dyscrasias, etc...
9. Any clinically significant moderate to severe sensory deficit lasting greater than 30 days after the first Exablate thalamotomy NOTE: Subjects with clinically significant moderate to severe sensory deficit following first Exablate thalamatomy should be excluded even if event resolves within a few months of treatment. This may cause new first thalamotomy subjects to be ineligible for the bilaterally staged treatment.
10. Moderate to severe cerebellar disturbance (imbalance or ataxia) or presence of moderate or severe hemiparesis NOTE: Subjects with moderate to severe cerebellar disturbance (imbalance or ataxia) or presence of moderate or severe hemiparesis following first Exablate thalamatomy should be excluded even if event resolves within a few months of treatment. This may cause new first thalamotomy subjects to be ineligible for the bilaterally staged treatment.
11. Any persistent dysphasia/dysarthria, language impairment following first Exablate thalamotomy.

    NOTE: Subjects with significant impairment following first Exablate thalamotomy should be excluded even if event resolves within a few months of treatment. This may cause new first thalamotomy subjects to be ineligible for the bilaterally staged treatment.
12. Significant reduction in cognitive function since the first thalamotomy. NOTE: Subjects with significant reduction in cognitive function following first Exablate thalamatomy should also be excluded even if event resolves within a few months of treatment. This may cause new first thalamotomy subjects to be not eligible for the bilaterally staged treatment.
13. Subject is pregnant or breastfeeding.
14. Subjects who have an overall Skull Density Ratio of less than 0.40 as calculated at screening

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Clinical Rating Scale for Tremor (CRST) | Baseline through Month 12 after First and Second Treatment
  The CRST is a standard tremor rating scale which measures subjects' tremor (Part A), motor Function (Part B), and Activities of Daily Living (Part C). Scores range from 0-4 with 0 being no tremor.
Incidence of Device and Procedure related Adverse Events | Treatment through Month 12 after Second Treatment
  All AEs will be reported and categorized by investigators in relation to the device or procedure, disease or unrelated to the device or procedures and categorized by first or second Exablate thalamotomy.

CONTACTS AND LOCATIONS:
Locations (2):
- HM CINAC, Móstoles, Madrid, Spain
- Imperial College, London, United Kingdom